CLINICAL TRIAL: NCT06306417
Title: Department of Traditional Chinese Medicine (TCM), Center for Reproductive Medicine, Department of Obstetrics and Gynaecology, Peking University Third Hospital, Beijing 100191, China.
Brief Title: A Randomized Controlled Trial of Acupuncture for Insulin Resistance in Patients With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKUTH TCM
Record Dates: First submitted 2024-02-19; First posted 2024-03-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-01

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): acupuncture
  Interventions: Other: lifestyle intervention; Device: acupuncture
- control group (Sham Comparator): sham acupuncture
  Interventions: Other: lifestyle intervention; Device: Sham acupuncture

INTERVENTIONS:
Other: lifestyle intervention — lifestyle intervention
Device: acupuncture — acupuncture
  Arms: Experimental group
Device: Sham acupuncture — Sham acupuncture
  Arms: control group

SUMMARY:
To determine the efficacy and safety of 2 different treatment modalities: 1) acupuncture plus lifestyle management (treatment group), 2) placebo plus lifestyle management (control group) in the treatment of insulin resistance in PCOS patients.

DETAILED DESCRIPTION:
A prospective, randomized controlled trial design was used to select women with polycystic ovary syndrome as the research subjects. 144 subjects who met the inclusion and exclusion criteria were randomly divided into an acupuncture plus lifestyle intervention group (treatment group) and a placebo plus lifestyle intervention group (control group). The differences in glucose metabolism and reproductive endocrinology were compared between the two groups.

1. To verify the efficacy and safety of acupuncture intervention on insulin resistance in PCOS;
2. To explore the effects of acupuncture on androgen and lipid levels, ovarian function, reproductive dysfunction, mood and quality of life in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* For the PCOS group, PCOS diagnosis according to Rotterdam criteria 2003 with at least two of the following three symptoms: (1) infrequent ovulation or anovulation; (2) hyperandrogenism or clinical manifestations of high blood androgen; (3) ultrasound findings of polycystic ovaries in 1 or 2 ovaries, or ≥12 follicles measuring 2 to 9 mm in diameter, and/or ovarian volume ≥10 mL

Exclusion Criteria:

1. Exclusion of other endocrine disorders such as androgen secreting tumors, suspected Cushing's syndrome and non-classic congenital adrenal hyperplasia (17-hydroxyprogesterone < 3nmol/L) thyroid dysfunction and hyperprolactinemia.
2. Type I diabetes or not well controlled type II diabetes
3. Stage 2 hypertension (resting blood pressure ≥160/100mmHg)
4. Psychiatric diagnoses or using psychiatric medications including antidepressants
5. Pharmacological treatment (cortizone, antidepressant, other antidiabetic treatment such as insulin and acarbose, hormonal contraceptives, hormonal ovulation induction or other drugs judged by discretion of investigator) within 12 weeks. Depo Provera or similar within 6 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | baseline and after 4 months
  calculation of HOMA-IR: [fasting insulin (μU/mL) × fasting glucose (mmol/L)] / 22.5)
  [Time Frame: Baseline]

SECONDARY OUTCOMES:
Hirsutism(FG score >4）, acne and early alopecia | baseline and after 4 months
  general condition
AUC insulin | baseline and after 4 months
  during oral glucose tolerance test (OGTT), AUCarea under the glucose tolerance curve
Follicle stimulating hormone (FSH) | baseline and after 4 months
  Examined with the blood sample
luteinizing hormone (LH) | baseline and after 4 months
  Examined with the blood sample
Progestin (P) | baseline and after 4 months
  Examined with the blood sample
Estrogen (E2) | baseline and after 4 months
  Examined with the blood sample
Prolactin (PRL) | baseline and after 4 months
  Examined with the blood sample
Androgen(T) | baseline and after 4 months
  Examined with the blood sample
Anti-mullerian hormone (AMH) | baseline and after 4 months
  Examined with the blood sample
Sex hormone-binding globulin (SHBG) | baseline and after 4 months
  Examined with the blood sample
Free testosterone index (FAI) | baseline and after treatment
  testosterone (nmol/ml) ×100 / SHBG (nmol/ml).
total cholesterol | baseline and after 4 months
  Examined with the blood sample
triglycerides | baseline and after 4 months
  Examined with the blood sample
high density lipoprotein (HDL) | baseline and after 4 months
  Examined with the blood sample
low density lipoprotein (LDL) | baseline and after 4 months
  Examined with the blood sample
Bile acidomics | baseline and after 4 months
  Quantitative detection of bile acids in blood and feces by targeted metabolomics (ultra-performance liquid chromatography-time-of-flight mass spectrometry).
Metagenomics and 16S rDNA sequencing analysis | baseline and after 4 months
  gDNA was extracted by fecal genomic DNA kit and sequenced by Illumina Hiseq 4000.
short form-36 (SF36) | baseline and after 4 months
  determine the health quality of life by the questionnaire of SF36 (0-100 score), the higher, the better
Self-Rating Anxiety Scale (SAS) | baseline and after 4 months
  determine the anxiety level with the questionnaire of SAS (20-100 score), the higher, the worse.
Self-Rating Depress Scale (SDS) | baseline and after 4 months
  determine the depress level with the questionnaire of SDS (20-100 score), the higher, the worse
polycystic ovary syndrome questionnaire, PCOSQ | baseline and after 4 months
  Mood, weight, body hair, acne, infertility, menstrual symptoms, and menstrual predictability in women with PCOS
BMI | baseline and after 4 months
  calculation:BMI=weight(kg)/height(m)^2
Fat% | baseline and after 4 months
  examined by body composition analyzer
waist to hip ratio(WHR) | baseline and after 4 months
  calculation of WHR: waist circumference(cm)/ hip circumference(cm)
glycosylated hemoglobin level | baseline and after 4 months
  Examined with the blood sample
ovarian size | baseline and after 4 months
  baseline and after 4 months, explained by 3 diameters: length(cm) * width(cm) * height(cm)
number of follicles | baseline and after 4 months
  observed by B-ultrasound
uterine size | baseline and after 4 months
  observed by B-ultrasound
endometrial thickness | baseline and after 4 months
  observed by B-ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Haolin Zhang, Study Director — Peking University Third Hospital
Locations (1):
- Peking University third hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
We haven't decided whether to share the data